CLINICAL TRIAL: NCT01846728
Title: Ovarian Function and Facultative Thermogenesis
Brief Title: Effects of Estrogen Deficiency on Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13-0149; P50HD073063 (NIH)
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Estrogen suppression (Experimental): Estrogen production will be suppressed using Lupron, a drug that blocks normal production of ovarian hormones
  Interventions: Drug: Estrogen suppression

INTERVENTIONS:
Drug: Estrogen suppression — Estrogen production will be suppressed for 3 months by administering a drug, lupron, that suppresses ovarian function
  Other Names: Lupron

SUMMARY:
Menopause is associated with weight gain, but the reasons why are not clear. In this study, the investigators will determine if reducing estrogen levels causes a decrease in the ability of the body to produce heat. If so, this would suggest this is one way that menopause may cause weight gain.

DETAILED DESCRIPTION:
The purpose of this pilot study is to investigate the role of the female sex hormone estrogen, on metabolism, thermoregulation and energy expenditure. Weight and fat gain increase after the menopause, but reasons for this are not clear. Loss of estrogen may cause changes in how women regulate metabolism and thermoregulation, possibly leading to weight gain. Specifically, this study will determine how loss of estrogen affects facultative thermogenesis. Loosely defined, facultative thermogenesis represents heat production that is turned on when needed. For example, when body core temperature falls below a certain threshold, a shivering response is invoked in skeletal muscle to increase heat production and, thus, energy expenditure. However, exposure over several hours to mild cold temperatures that do not trigger shivering (16-20⁰ C) also induces an increase in energy expenditure (cold-induced non-shivering thermogenesis). Although several different tissues may contribute to this response, the recent identification of functional brown adipose tissue (BAT) in humans has promoted an interest in how BAT is activated in humans and its potential role in regulating energy balance and body weight. The investigators will measure BAT activity using PET/CT scans pre and post three months of estrogen suppression.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index < 30 kg/m2
* Normal menstrual cycles
* Premenopausal

Exclusion Criteria:

* irregular menstrual cycles defined as 2 or more missed cycles in the previous year
* on hormonal contraceptive or menopausal therapy
* positive pregnancy test
* intention to become pregnant or start hormonal contraceptive therapy during the period of study
* lactation
* severe osteopenia or osteoporosis (i.e., proximal femur or lumbar spine t scores < -2.0)
* abnormal vaginal bleeding
* thyroid dysfunction
* uncontrolled hypertension
* exercising at least 30 minutes per day at a moderate to vigorous intensity >1 d/wk) over the past 6 months

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-04; Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Melanson, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through advertisements posted on the Anschutz Medical Campus and distributed through the campus email system. 12 women consented to participate in the study (consent was obtained prior to screening and orientation). After the screening and orientation process, 6 elected to continue, and 6 elected not to continue
Groups:
- Estrogen Suppression: Estrogen production will be suppressed using Lupron, a drug that blocks normal production of ovarian hormones
  Estrogen suppression: Participants underwent 3 mo of ovarian hormone suppression using the GnRHAG leuprolide acetate (Lupron; TAP Pharmaceutical Products, Inc; Lake Forest, IL) delivered by monthly intramuscular injection (3.75 mg).
Period: Overall Study
Arm/Group | Estrogen Suppression
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Estrogen Suppression
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.3 (4.5)
Weight [Mean (Standard Deviation); unit: kg] | 64.8 (16.3)
Fat mass (measured with DXA) [Mean (Standard Deviation); unit: kg] | 24.2 (8.9)
fat free mass (from DXA) [Mean (Standard Deviation); unit: kg] | 40.3 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Brown Adipose Tissue Activity
Description: Brown adipose tissue activity will be measured using Positron Emission Tomography/computer tomography (PET/CT) before and after 3 months of estrogen suppression. Activity is quantified as the standard uptake value (SUV), It is a mathematically derived ratio that is a semiquantitative measure of the tracer uptake in a region of interest that normalizes the lesion activity to the injected activity and a measure of the volume of distribution (usually total body weight or lean body mass).
Time Frame: Baseline and after 3 months of suppression
Measure: Mean (Standard Deviation); unit: Standard uptake value (SUV)
Arm/Group | Estrogen Suppression
Number analyzed (Participants) | 6
Standard uptake value (SUV)
  Baseline | 3.9 (1.8)
  3 mo | 4.0 (2.0)
Statistical Analysis 1: Comparison: Estrogen Suppression; Test type: Other; p = 0.84, t-test, 2 sided — Because this was a pilot study, the study was not powered to detect differences over time. the study was performed to generate preliminary data on means and standard deviations

2. Secondary Outcome: Cold Induced Thermogenesis
Description: The increase in energy expenditure above resting during cold exposure
Time Frame: Baseline and after 3 months of suppression
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Estrogen Suppression
Number analyzed (Participants) | 6
kcal
  Baseline | 350 (228)
  3 mo | 301 (139)
Statistical Analysis 1: Comparison: Estrogen Suppression; Because this was a pilot study, the study was not powered to detect differences over time. the study was performed to generate preliminary data on means and standard deviations; Test type: Other; p = 0.66, t-test, 2 sided

3. Secondary Outcome: Fat Mass
Description: Amount of body fat (in kg)
Time Frame: Baseline and after 3 months of suppression
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Estrogen Suppression
Number analyzed (Participants) | 6
kg
  Baseline | 24.2 (8.9)
  3 mo | 24.1 (4.5)
Statistical Analysis 1: Comparison: Estrogen Suppression; Test type: Other — Because this was a pilot study, the study was not powered to detect differences over time. the study was performed to generate preliminary data on means and standard deviations; p = 0.92, t-test, 2 sided

4. Secondary Outcome: Fat Free Mass
Description: Fat free mass measured by DXA
Time Frame: Baseline and after 3 mo of suppression
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Estrogen Suppression
Number analyzed (Participants) | 6
kg
  Baseline | 40.3 (8.4)
  3 mo | 40.4 (8.3)
Statistical Analysis 1: Comparison: Estrogen Suppression; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.98, t-test, 2 sided

5. Secondary Outcome: Resting Energy Expenditure
Description: Energy expenditure measured in the resting state
Time Frame: after 3 months of suppression
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Estrogen Suppression
Number analyzed (Participants) | 6
kcal
  Baseline | 1382 (218)
  3 mo | 1340 (209)
Statistical Analysis 1: Comparison: Estrogen Suppression; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.66, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Estrogen Suppression
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estrogen Suppression (N=6)
Vaginal Bleeding (Reproductive system and breast disorders) | 1 (1)
Headaches (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a pilot study to generate preliminary data for an NIH grant application. there was insufficient power to detect significant differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No